CLINICAL TRIAL: NCT01365234
Title: Model 20066 Left Ventricular (LV) Lead Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Model 20066
Record Dates: First submitted 2011-05-25; First posted 2011-06-03 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20066 Lead (Experimental): Non-randomized study. Intervention: Device: Pacing Lead
  Interventions: Device: Pacing Lead

INTERVENTIONS:
Device: Pacing Lead — Implant and follow up of Model 20066 lead

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. When there are changes in the heart beat sometimes an implantable heart device is used to control the rate and rhythm of the heart beat. In certain heart failure cases, when the two lower chambers of the heart no longer beat in a coordinated manner, cardiac resynchronization therapy (CRT) may be prescribed. CRT is similar to a pacemaker. It is placed (implanted) under the skin of the upper chest. CRT is delivered as tiny electrical pulses to the right and left ventricles through three leads (flexible insulated wires) that are inserted through the veins to the heart. The purpose of this study is to evaluate a new lead for delivering energy to the left ventricle (bottom left chamber of the heart).

ELIGIBILITY:
Inclusion Criteria:

* Patient meets CRT inclusion criteria as determined by local regulatory and/or hospital policy
* Patient has signed and dated the study-specific informed consent form
* Patient is 18 years of age or older
* Patient is expected to remain available for follow-ups at the investigational center
* Patient is willing and able to comply with protocol

Exclusion Criteria:

* Patient has a previous complete atrial based biventricular CRT system
* Patient has a previous LV lead implanted or previous implant attempt within 30 days of implant or ongoing Adverse Events from previous unsuccessful attempt
* Patient has known coronary venous vasculature that is inadequate for lead placement
* Patient has unstable angina pectoris or has had an acute myocardial infarction (MI) within the past month
* Patient has had a coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within the past three months
* Patient has chronic (permanent) atrial arrhythmias
* Patient has contraindications for standard transvenous cardiac pacing (e.g., mechanical right heart valve)
* Patient has had a heart transplant (patients waiting for heart transplants are allowed in the study)
* Patient is enrolled in any concurrent drug and/or device study that may confound the results of this study
* Patient has a terminal illness and is not expected to survive more than three months
* Patient meets exclusion criteria required by local law (e.g. age, incompetence, pregnancy, breast feeding, etc).
* Patient is unable to tolerate an urgent thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of implant procedure related and lead-related complications in the first month post-implant | One Month

SECONDARY OUTCOMES:
Success rate of the Model 20066 lead | Within 24 hours of procedure initiation
Cannulation time | Within 24 hours of procedure initiation
Fluoroscopy Time | Within 24 hours of procedure initiation
Model 20066 Lead Placement Time | Within 24 hours of procedure initiation
Total Implant Time | Within 24 hours of procedure initiation
Assessment of Lead Handling Characteristics | Within 24 hours of procedure initiation
Electrical Performance-Tip Electrode: LV Voltage Threshold | 12-month
Electrical Performance -Tip Electrode: Sensing | 12-month
Electrical Performance -Tip Electrode: Pacing Impedance | 12-month
Electrical Performance -Ring Electrode: LV Voltage Threshold | 12-month
Electrical Performance -Ring Electrode: Sensing | Within 24 hours of procedure initiation
Electrical Performance -Ring Electrode: Pacing Impedance | 12-month
Summarize All Adverse Events | 12-month
Summarize Final 20066 Lead Position | Within 24 hours of procedure initiation

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Yee, MD, Principal Investigator — London Health Sciences Centre, London, Ontario, Canada
Locations (4):
- Canada (2):
  - London
  - Newmarket
- Kuala Lumpur, Malaysia
- Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yee R, Gadler F, Hussin A, Bin Omar R, Khaykin Y, Verma A, Lazeroms M, Hine DS, Marquard KR. Novel active fixation mechanism permits precise placement of a left ventricular lead: early results from a multicenter clinical study. Heart Rhythm. 2014 Jul;11(7):1150-5. doi: 10.1016/j.hrthm.2014.04.020. Epub 2014 May 4. PMID 24801899